CLINICAL TRIAL: NCT07151846
Title: Discovery and Validation of Digital Phenotypes for Predicting Recurrence of Depressive Episodes
Brief Title: Digital Phenotypes for Predicting Depression
Status: Enrolling by invitation | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Korea University Medicine (Unknown); Hucircadian (Industry)
Responsible Party: Principal Investigator, Heon-Jeong Lee, MD, PhD, Professor, Korea University Anam Hospital
Other Study IDs: MY MENTAL HERO; RS-2024-00469788 (Other: National Research Foundation of Korea (NRF))
Record Dates: First submitted 2025-07-23; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Depression - Major Depressive Disorder; Depression Bipolar; Bipolar Disorder (BD); Mood Disorders
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient group: Adults (19-75 years) with a clinical diagnosis of a major mood disorder (bipolar I/II or major depressive disorder) per DSM-5, with at least one prior depressive episode.
- High Risk: Adults (19-75 years) with no formal diagnosis of bipolar disorder or major depressive disorder, but who meet at least one of the following:
  1. Elevated scores at screening (K-MDQ ≥7 or PHQ-9 ≥5), or
  2. Report of persistent mood symptoms (e.g., ≥2 weeks of low mood or ≥several days of elevated/irritable mood) during MINI interview.
- Healthy Control: Adults (19-75 years) with no current or past diagnosis of bipolar disorder or major depressive disorder, and who screen below cutoff on both K-MDQ (<7) and PHQ-9 (<5).

SUMMARY:
This longitudinal study aims to identify and validate digital phenotypes that can predict recurrence of major depressive episodes using passively collected, real-time sensing data from smartphones and wearable devices. Over a 12-month period, 540 participants-including patients with mood disorders and healthy or high-risk controls-will complete five clinical assessments at 3-month intervals, wear a Fitbit device daily, and log daily mood ratings via a mobile app. The study includes the development of AI-based predictive models and the construction of an anonymized wearable big-data repository for mood disorders.

DETAILED DESCRIPTION:
This is a 12-month longitudinal follow-up study designed to identify digital phenotypes capable of predicting the recurrence of major depressive episodes using passively collected real-time data from smartphones and wearable devices. A total of 540 participants will be enrolled, including 200 patients diagnosed with mood disorders who have experienced at least one depressive episode in the past two years, and 340 healthy or high-risk control participants without a clinical diagnosis.

Clinical interviews and self-report measures will be conducted five times at 3-month intervals. Throughout the study period, participants will wear a Fitbit device daily and use the "My Mental Hero" mobile application to record their mood once a day at a self-selected time. Data collected will be used to develop machine learning models for predicting depressive recurrence and to build a large-scale, anonymized wearable big-data repository for mood disorders.

Participants will receive no interventions beyond data collection, and neither randomization nor blinding will be implemented. Trained psychiatrists, clinical psychologists, or research nurses will conduct the assessments. Initial visits will include informed consent, device setup, and app training, taking approximately 1-2 hours. Subsequent assessments will take about one hour, with additional brief interviews (≤30 minutes) conducted if a mood episode is suspected.

While follow-up assessments for patients and high-risk participants will be conducted in person, those for healthy controls may be conducted remotely (via Zoom or phone) under secure and private conditions without screen recording. Remote assessments may also be used for patient and high-risk groups if necessary.

ELIGIBILITY:
Inclusion Criteria for Patient Group:

1. Adults aged 19 to 75 years and 11 months.
2. Diagnosed with a major mood disorder (bipolar I or II disorder, or major depressive disorder) based on DSM-5, with a history of psychiatric visits for mood symptoms.
3. Has experienced at least one prior depressive episode (major, minor, or brief).
4. Owns a smartphone with stable internet connectivity, can operate it without difficulty, and agrees to install a digital phenotyping application, wear a Fitbit device daily, and complete daily mood logs throughout the study period.

Inclusion Criteria for Healthy Control Group:

1. Adults aged 19 to 75 years and 11 months.
2. No current or past diagnosis of bipolar disorder or major depressive disorder.
3. Scores below clinical thresholds on both K-MDQ (<7) and PHQ-9 (<5) at baseline assessment.
4. Owns a smartphone with stable internet connectivity, can operate it without difficulty, and agrees to install a digital phenotyping application, wear a Fitbit device daily, and complete daily mood logs throughout the study period.

Inclusion Criteria for Hight Risk Group:

1. Adults aged 19 to 75 years and 11 months.
2. No current or past diagnosis of bipolar disorder or major depressive disorder.
3. Meets either of the following:

   A. Scores above the threshold on K-MDQ (≥7) or PHQ-9 (≥5) at baseline. B. Reports persistent mood symptoms during MINI (e.g., ≥2 weeks of depressive mood/anhedonia, or several days of elevated/irritable mood).
4. Owns a smartphone with stable internet connectivity, can operate it without difficulty, and agrees to install a digital phenotyping application, wear a Fitbit device daily, and complete daily mood logs throughout the study period.

Exclusion Critera (Overall)

1. Inability to provide informed consent due to cognitive impairment, severe psychiatric symptoms, or language barriers.
2. Presence of any neurological or medical condition that may significantly affect mood, cognition, or behavior (e.g., epilepsy, dementia, traumatic brain injury).
3. Current substance use disorder or dependence (excluding nicotine or caffeine) that is either untreated or clinically unstable.
4. Severe suicidal ideation or risk as determined by clinical judgment at screening.
5. Ongoing participation in another interventional clinical trial, particularly those involving psychotropic medications or digital health interventions.
6. Inability or unwillingness to wear a wearable device (Fitbit) or use the required mobile application daily throughout the study.
7. Lack of stable internet access or a compatible smartphone required for digital phenotyping data collection.
8. Any other condition that, in the investigator's judgment, may compromise the participant's safety, compliance, or the integrity of the study data.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit a total of 540 participants divided into three groups:
  Patient Group (PT, n=200):
  Individuals diagnosed with a mood disorder (bipolar I/II or major depressive disorder) who have experienced at least one depressive episode within the past two years.
  High-Risk Group (HR):
  Individuals with no formal mood disorder diagnosis but who present subclinical mood symptoms or elevated screening scores suggesting potential risk for affective disorders.
  Healthy Control Group (HC):
  Individuals with no history or current diagnosis of any mood disorder and who do not show clinically significant symptoms on screening assessments.
  All participants will undergo 5 clinical assessments over a 12-month period (every 3 months) and will be asked to wear a Fitbit device daily and record their mood daily via a mobile app throughout the study. No therapeutic intervention will be provided, and the study does not involve randomization or blinding.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The Patient Health Questionnaire (PHQ-9) | Baseline, month 3, month 6, month 9, month 12
  The Patient Health Questionnaire (PHQ-9) is a self-report screening tool designed to assess the severity of depressive symptoms. PHQ score range is 0 to 27. Higher PHQ score indicates worse depressive symptoms.
Inter-visit mood episode occurance | month 3, month 6, month 9, month 12
  Mood episodes that occur between scheduled study visits will be assessed by trained raters. If an inter-visit episode is suspected, a structured clinical evaluation will be conducted using standardized case report forms (CRFs) to determine:
  1. Episode period (start and end dates),
  2. Presence of DSM-5 mood symptoms (e.g., depressed mood, anhedonia, decreased need for sleep, inflated self-esteem),
  3. Episode severity as rated by the Clinical Global Impressions (CGI) scale (1-7; higher scores indicate greater severity).
  Scoring and Interpretation:
  * CGI scale range: 1 (Normal, not ill) to 7 (Among the most extremely ill patients).
  * Higher CGI scores represent worse mood symptom severity.
  Diagnostic criteria for depressive episodes (≥1 core symptom plus ≥5 symptoms, ≥2 weeks) and (hypo)manic episodes (≥1 core symptom plus ≥3-4 symptoms, ≥4 days) will be applied using the CRF.
MADRS (Montgomery-Åsberg Depression Rating Scale) | Baseline, month 3, month 6, month 9, month 12
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-administered tool used to assess the severity of depressive symptoms. It consists of 10 items rated on a 0-6 scale and is widely used in clinical trials due to its sensitivity to treatment-related change. MADRS score range is 0 to 60. Higher MADRS score indicates worse depressive symptoms.
YMRS (Young Mania Rating Scale) | Baseline, month 3, month 6, month 9, month 12
  The Young Mania Rating Scale (YMRS) is a clinician-rated scale used to measure the severity of manic symptoms in individuals with bipolar disorder. It includes 11 items covering mood, behavior, and cognitive functioning, with higher scores indicating greater symptom severity. YMRS score rang is 0 to 60.
  Higher YMRS score indicates worse manic symptoms.
CGI (Clinical Global Impression Scale) | Baseline, month 3, month 6, month 9, month 12
  The Clinical Global Impression (CGI) Scale is a standardized assessment tool used by clinicians to rate overall illness severity (CGI-S). CGI-S is rated on a 7-point scale for each of three components: Depression, Mania, Overall. CGI scale range: 1 (Normal, not ill) to 7 (Among the most extremely ill patients).

CONTACTS AND LOCATIONS:
Overall Officials: Heon-Jeong Lee, Professor, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, Seongbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Some of the data will be shared with the K-BDS (Korea Brain Data Station) after the completion of the study; however, the exact amount and timing of data to be shared have not yet been determined. The expected date of upload to the K-BDS is December 31, 2027.